CLINICAL TRIAL: NCT04488471
Title: Impact of Isolation in Patients With IBD During the 2020 COVID-19 Crisis: a Mixed Methods Study
Brief Title: Impact of Isolation in Patients With IBD During the COVID-19 Crisis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH21414
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- high-risk group: IBD patients who were high risk of infection and were shielding
- low-risk group: IBD patients who were low risk of infection and were following standard quarantine guidance
- young people from affiliated study: 32 IBD patients from an affiliated study

SUMMARY:
The coronavirus pandemic has changed healthcare dramatically in a short time. Individuals with chronic illnesses and services for them have had to adapt and change to deal with requirements for shielding and social isolation to reduce infection risk and management of medication investigation and ongoing review.

It is increasingly recognised that the pandemic and the changes to daily life will have had a series of impacts on patients and health care services, including impacts on patients psychological well-being and the opportunity to seek medical care for non-CoViD illness.

Psychological symptoms such as depression, anxiety and hopelessness is well described in adults and young people with inflammatory bowel disease. Quarantine has also been associated with these psychological symptoms and also post-traumatic stress. It is important to identify the extent of and factors that influence negative psychological consequences of isolation in patients with inflammatory bowel disease.

This study will aim to assess what impact the isolation of patients during social isolation had in terms of psychological well-being - and what are the factors affecting this impact, particularly in younger and old age groups.

DETAILED DESCRIPTION:
This study will use both questionnaires and semi-structured interviews to understand how IBD patients have been impacted psychologically by the CoViD-19 pandemic and identify various factors that may affect the extent to which patients have been impacted. This study will also incorporate longitudinal questionnaire follow-up of the same patients, in order to try and understand the long-term impact of the pandemic, and to assess changes in psychological impact accompanying changes in the national situation.

Patients identified from those attending the IBD clinic will be contacted. As part of the NHSE and local Trust CoViD response, lists of all patients attending the IBD clinics and those deemed to be at high risk of infection have been created.

This study aims to recruit 100 patients from the high-risk group and 100 patients from the non-high-risk group. Basedon an approximately 33% response rate, we have therefore elected to identify 300 patients from the high-risk groups and 300 from non-high-risk groups. These 600 patients in total will be contacted via the post, and mailed:

1. An explanatory cover letter, with instructions on how to participate in the study
2. Participant information sheet (PIS)
3. Consent form
4. Questionnaires
5. A stamped and addressed return envelope

Completion of questionnaire and return to site will constitute as consent for this data to be used. Postal recruitment is being used to maximise the chances of reaching those who may have been most affected by isolation and may have limited access to the internet. The consent form will apply to the optional interview component.

The PIS will include information signposting patients to help and support should they have difficulties or concerns relating to the study or the psychological impact of their condition or current situation.

Record of who has been contacted to participate will be kept on NHS computers, with patient hospital numbers corresponding to anonymous and non-identifiable study identification numbers. Keeping record will permit there to be available data regarding the questionnaire return rate. This will also potentially allow for demographic details to be retrieved from patient records regarding those who did not return responses, to facilitate both assessment of differences between responders and non-responders and provide information about those who elected not to participate.

In addition, a sub-set of 32 young people will be contacted and recruited. This sub-set have already undertaken the assessment of psychological morbidity, outlined below, during a previous, pre-CoViD outbreak study (STH20960 IRAS: 269881) and have agreed to further follow-up. These patients will also be contacted via the post to complete the same set of questionnaires and therefore provide follow-up, to assess whether measures of psychological morbidity changed following the onset of the CoViD crisis.

Patients will be asked to complete the following questionnaires:

1. IBD symptoms: IBD control questionnaire
2. Experience during the CoViD periods of isolation
3. Impact of event scale (iES-15 questionnaire)
4. Depression Anxiety Stress Scale-21 (DASS-21)

Background information, as listed below, will be collected in order to try and identify demographic and disease related details which may affect the level of psychological impact for IBD patients:

1. Age
2. Ethnicity
3. Postcode (used to calculate indices of deprivation scores, using the Indices of Multiple Deprivation [IMD] tool)
4. Disease type
5. Medication
6. BSG risk group

The same patients will be contacted and asked to complete the questionnaires again after 6 and 12 months to assess changes in psychological impact and relationship to societal requirements for isolation.

Semi structured interviews will be undertaken with approximately 20 participants. More may be undertaken until saturation point is reached.

Semi-structured interviews will be undertaken to provide further detail about the experience of isolation during the pandemic to explore issues to include factors which improve or worsen the experience of isolation including:

* The effect of the isolation itself
* The effect of variations in information provision
* Concern about infection risk and its variation during the period of "lock-down"
* Delays to presentation with flare symptoms

ELIGIBILITY:
Inclusion Criteria:

* IBD Patients who utilise the IBD Clinics at Sheffield Teaching Hospitals NHS FT

Exclusion Criteria:

* patients who are not part of the IBD clinics at STH NHS FT

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a clinical diagnosis of IBD who are treated in the clinics of Sheffield Teaching Hosptials NHS FT
Sampling Method: Non-Probability Sample
Enrollment: 232 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
What impact has the isolation of patients during social isolation had in terms of psychological morbidity? | Changes in psychological morbidity at 12 months
  Psychological morbidity will be assessed through the 4 questionnaires

SECONDARY OUTCOMES:
Have levels of psychological morbidity in young people changed from levels prior to the CoViD pandemic? | Changes in psychological morbidity at 12 months
  psychological morbidity will be assessed via comparison of questionnaires from affiliated study against the time points of this study

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lobo, MD, Study Chair — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Sheffield Teaching Hospitals NHS FT, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no IPD will be shared with other researchers